CLINICAL TRIAL: NCT06246864
Title: Evaluation of the Effects on the Skin of Different Materials Used in Orogastric Tube Detection in Premature Babies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra TURAL BUYUK, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Flaster
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Skin Conditions
Keywords: premature; skin care; Hydrocolloid dressing; hypoallergenic patch
MeSH Terms: conditions — Premature Birth | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: randomized control experimental trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocolloid dressing group (Experimental): The premature baby's Oragastric tube will be fixed using a hydrocollaid dressing. Orogastric fixation will not be changed for 24 days. After 24 hours, the fixed patch will be removed using a silicone-based spray remover.
  Interventions: Other: Hydrocolloid dressing
- Hypoallergenic Flexible Patch group (Active Comparator): Oragastric tube of premature baby Hypoallergenic Flexible Patch will be detected using . Orogastric fixation will not be changed for 24 days. After 24 hours, the fixed patch will be removed using a silicone-based spray remover.
  Interventions: Other: Hypoallergenic Flexible

INTERVENTIONS:
Other: Hydrocolloid dressing — After the oral gastric tube is placed on the premature baby and fixed with a Hydrocolloid dressing, the fixed patch will be removed after 24 hours using a silicone-based spray remover.
  Arms: Hydrocolloid dressing group
Other: Hypoallergenic Flexible — After the oral gastric tube is placed on the premature baby and fixed with a hypoallergenic flexible patch, the fixed patch will be removed after 24 hours using a silicone-based spray remover.
  Arms: Hypoallergenic Flexible Patch group

SUMMARY:
While medical adhesives provide fixation of devices and catheters in neonatal intensive care, they can cause disruption of skin integrity when removed. Therefore, when detecting medical devices, it is important to choose products that will not harm babies' skin and to use different occlusive dressings (polymer foams, hydrogel dressings, hydrocolloid dressings).

This study aims to compare the effectiveness of different types of patches (Hydrocolloid dressing and Hypoallergenic Flexible Patch) used in the detection of oragastric catheter (OG) in preterm babies hospitalized in the neonatal intensive care unit in preventing skin damage.

DETAILED DESCRIPTION:
Many interventions are applied to premature babies in neonatal intensive care units due to the developing technologies in recent years. Babies in neonatal intensive care need many devices to maintain their vital functions and monitor the treatment process. The medical adhesive materials to be selected are important in determining the medical devices used in neonatal intensive care units, especially premature babies.

This study aims to compare the effectiveness of different types of patches (Hydrocolloid dressing and Hypoallergenic Flexible Patch) used in the detection of oragastric catheter (OG) in preterm babies hospitalized in the neonatal intensive care unit in preventing skin damage.

ELIGIBILITY:
Inclusion Criteria:

* A newborn is a baby born between 32-36 weeks of gestation
* No medical adhesive tape should be applied to the newborn's lips beforehand.
* The newborn does not have any skin diseases
* OG will be inserted into the newborn for the first time
* Having a newborn receiving respiratory support with non-invasive mechanical ventilation, hood or free oxygen

Exclusion Criteria:

* The newborn is not a baby born between 32-36 weeks of gestation
* Applying medical adhesive tape on the newborn's lips beforehand
* The newborn has any skin disease
* OG has been inserted into the newborn before and detected.
* Supporting and detecting the newborn's breathing by intubating it

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Newborn Skin Condition Score | The patch will be removed 24 hours after orogastric detection and a skin evaluation will be performed immediately.
  NSCS allows evaluation of the newborn's skin condition. It evaluates skin dryness, redness and integrity, which are the basic characteristics of the newborn's skin. The scale consists of three parameters.

IPD SHARING:
Plan to Share IPD: No